CLINICAL TRIAL: NCT02989571
Title: A Double-Blinded Randomized Controlled Trial on the Effects of Increased Intravenous Hydration on Nulliparous Women Undergoing an Induction of Labor
Brief Title: The Effects of Increased IV Hydration on Nulliparous Women Undergoing an Induction of Labor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Principal Investigator, Vineet Shrivastava, Principal Investigator, MemorialCare Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 628-15
Record Dates: First submitted 2016-01-21; First posted 2016-12-12 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Labor; Forced or Induced, Affecting Fetus or Newborn
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: A power size calculation was performed using previously published institutional data as well as previously reported literature regarding induction of labor in nulliparous women. Baseline duration of labor induction among nulliparous women range from 21-30 hours. In order to obtain 80% power to detect a 20% decrease in the duration of labor at a statistical significance level of 0.05, 73 participants are needed in each group. In order to account for participant withdrawal and enrollment errors, the sample size is increased to 90 per group for a total of 180 participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Placebo Arm (Placebo Comparator): Intravenous normal saline administered at 125ml/hr
  Interventions: Drug: Intravenous normal saline administered at 125ml/hr
- Group 2 - Intervention Arm (Active Comparator): Intravenous normal saline administered at 250ml/hr
  Interventions: Drug: Intravenous normal saline administered at 250ml/hr

INTERVENTIONS:
Drug: Intravenous normal saline administered at 250ml/hr — Intravenous normal saline administered at 250ml/hr
  Other Names: Normal saline
  Arms: Group 2 - Intervention Arm
Drug: Intravenous normal saline administered at 125ml/hr — Intravenous normal saline administered at 125ml/hr
  Other Names: Normal saline
  Arms: Group 1 - Placebo Arm

SUMMARY:
The objective of this study is to compare the effects of intravenous fluid rate on the course of labor in nulliparous patients who are undergoing labor induction and have an unfavorable cervix. The primary hypothesis is that an increased rate of intravenous fluids will shorten the length of labor in patients undergoing induction with an unfavorable cervix.

DETAILED DESCRIPTION:
Exercise physiology has shown that increased fluid intake and replacement can improve skeletal muscle performance in prolonged exercise. Labor is a physically demanding process that is essentially an "exercise" of the uterus, where uterine contractions of varying strength and dilation lead to thinning and dilation of the cervix and to eventual delivery of the infant. It has logically been theorized that, as with any exercise, improved hydration and delivery of carbohydrates to uterine smooth muscle can help optimize the contractions needed during labor. Conversely, dehydration is believed to result not only in decreased uterine perfusion (due to decreased intravascular volume), but also in reduced delivery of nutrients and elimination of waste products from the contracting myometrium.

Inadequate maternal hydration has been postulated to be a contributing factor to prolonged or dysfunctional labor, in which uterine contractions are not sufficiently strong or are inappropriately coordinated to cause adequate cervical dilation and effacement. Even in patients who completely dilate, sufficient voluntary and involuntary muscle effort is required during the second stage of labor to achieve a vaginal delivery. Prolonged labors can not only lead to increased hospitalization cost, but also to increased risks of cesarean delivery for indications such as "failure to progress," chorioamnionitis (intrauterine infection), and postpartum hemorrhage. Establishing techniques to optimize the length and duration of labor has therefore been an area of particular research interest.

To date, several randomized, controlled studies have demonstrated that with higher intravenous (IV) fluid rates, there is a decreased frequency of prolonged labor and possibly a decreased need for oxytocin in patients who present in active labor. One of these studies was performed here at Long Beach Memorial by Garite et al under IRB approval and supervision. Importantly, a systematic review of these studies by the Cochrane Collaboration in 2013 demonstrated that increased intravenous fluid rates (250mL/hr vs 125mL/hr) appears to shorten the time to delivery and the cesarean delivery rate in patients who present in active labor.

The rate of induction of labor has increased dramatically in recent years, from 9.5% in 1990 to 22.1% in 2004. Women undergoing an induction of labor (whether elective or medically indicated) represent a distinct population from those who present in active labor, not only with regards to their baseline characteristics, but also with regards to their labor course and maternal and neonatal outcomes. There have been no studies thus far investigating the use of increased intravenous hydration in patients undergoing induction of labor, as previous studies have focused on patients who present in active labor. The objective of this study is therefore to determine the effect of increased intravenous hydration in nulliparous patients undergoing an induction of labor on length of labor, mode of delivery, and other maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* ≥ 18 years of age
* Singleton gestation
* Nulliparous
* Vertex presentation
* Gestational age ≥ 36 weeks
* Bishop score ≤ 6
* undergoing induction of labor

Exclusion Criteria:

* Multiparous
* Preeclampsia at admission
* Gestational or chronic hypertension
* Non-vertex presentation
* Multiple gestation
* Chorioamnionitis at admission
* Intrauterine growth restriction (<10th percentile)
* BMI > 50
* Presence of uterine scar
* Participation in any other research protocol involving induction of labor
* Nonreassuring fetal heart rate tracing at admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Length of labor (hours of duration) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review

SECONDARY OUTCOMES:
Epidural use (yes or no) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
Oxytocin use (yes or no) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
Mode of Delivery (vaginal delivery, operative vaginal delivery, or cesarean) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
Indication for operative or cesarean delivery (e.g. Nonreassuring fetal tracing, arrest of labor, other) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
Maternal infectious or other morbidity (Yes or No) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
Birth weight (numerical value in grams) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
Neonatal weight at 72 hours of life (numerical value in grams) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
NICU admission (Yes or No) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
Need for treatment of jaundice (yes or no) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
NICU length of stay (numerical value expressed in days) | within the first 7 days (plus or minus 3 days) after delivery
  Measured via chart review
Delivery within 24 hours (yes or no) | within 24 hours after delivery
  Measured via chart review

CONTACTS AND LOCATIONS:
Overall Officials: Vineet Shrivastava, MD, Principal Investigator — Magella Medical Group
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: Undecided